CLINICAL TRIAL: NCT06253117
Title: Evaluation of Pirfenidone as a Novel Therapeutic Strategy Against Recurrent Acute Pancreatitis.
Acronym: PirfenidoneRAP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kondal Kyanam, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300012263; HT9425-23-1-0900 (Other Grant/Funding Number: DOD CDMRP)
Record Dates: First submitted 2024-01-20; First posted 2024-02-12 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Pirfenidone (Experimental): Pirfenidone Days 1-7: 267 mg PO TID (801 mg/day) Days 8-14: 534 mg PO TID (1602 mg/day) Day 15 and thereafter: 801 mg PO TID; not to exceed 2403 mg/day Total duration of experimental or placebo drug treatment 6 months
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone Days 1-7: 267 mg PO TID (801 mg/day) Days 8-14: 534 mg PO TID (1602 mg/day) Day 15 and thereafter: 801 mg PO TID; not to exceed 2403 mg/day
  Duration of treatment- total 6 months
  Arms: Pirfenidone
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This clinical will evaluate the safety, tolerability and early efficacy of pirenidone in patients with recurrent acute pancreatitis.

DETAILED DESCRIPTION:
Background: Recurrent Acute Pancreatitis (RAP) is occurrence of 2 or more distinct episodes of Acute Pancreatitis (AP) (separated by at least 3 months). RAP not only leads to significant morbidity and reduced quality of life; patients with RAP have a substantial (up to 40%) risk of progressing to chronic pancreatitis (CP). Unfortunately, there is no therapy, which can help prevent future attacks of pancreatitis in RAP patients. In this regard, our published work suggest that pirfenidone, a therapy approved by FDA for the treatment of Idiopathic Pulmonary Fibrosis (IPF), has the potential to emerge as a novel treatment for patients with RAP. Briefly, our results suggest that: 1) Pirfenidone, when administered prophylactically, reduces the risk of AP development; 2) Pirfenidone, when given to experimental animals with severe AP, leads to amelioration of local and systemic injury; and 3) Pirfenidone, when administered to experimental animals with ongoing RAP, reduces risk of progression to CP. Thus, our results suggest that pirfenidone has potential to emerge as novel therapeutic strategy for RAP patients. These studies have high translational value as pirfenidone is already in clinical use for IPF and has over 8 years of record of safety.

Hypothesis: "Pirfenidone treatment in patients with RAP will be safe, tolerable, and efficacious." Objectives: The study has following primary and secondary objectives. Primary Objective: 1) To evaluate the safety and tolerability of pirfenidone compared to placebo, in patients with RAP. 2) To evaluate the efficacy of pirfenidone in reducing the laboratory markers of inflammation.

Secondary Objective: 1) To evaluate the efficacy of pirfenidone in reducing- a) recurrence of AP; b) pancreatitis related emergency room visits and readmissions; c) severity of pancreatitis, if acute pancreatitis was to develop; d) Improving quality of life measures; e) Improvement in patient reported outcomes. 2) To develop a predictive biomarker of efficacy of pirfenidone, which can be incorporated in a future clinical trial.

Specific aims and study design. Pilot Clinical Trial of the Safety, Tolerability and Efficacy of Pirfenidone in RAP. We will conduct a randomized, double-blind, placebo controlled pilot trial of pirfenidone in patients with RAP. RAP patients, 18-85 years of age who meet the eligibility criteria, will be recruited at one of the three participating sites (UAB, Mayo clinic Rochester and Brigham and Women's Hospital, Boston), and randomly assigned to pirfenidone or placebo treatment for 6 months. The primary endpoints of this clinical trial are a) feasibility; and b) safety. We have multiple efficacy secondary endpoints endpoint like cumulative incidence and rate of recurrent attacks of AP, severity of recurrent attacks of AP (mild/moderate/severe), readmissions and/or ER visits for pain, changes in quality of life as measured by PANQOLI and SF-12 health survey questionnaires, and changes in changes in patient reported outcome as measured by PAN-PROMISE score. We plan to recruit 60 patients at the three study sites over the duration of this clinical trial.

ELIGIBILITY:
A- Inclusion Criteria:

1. Patients 18 - 85 years of age
2. Two or more documented attacks of acute pancreatitis, separated by 3 months from one another, defined by at least 2 of the following 3:

   1. amylase or lipase values, or both, that are greater than 3 times the upper limit of normal values
   2. characteristic cross-sectional imaging
   3. typical upper abdominal pain according to the revised Atlanta classification28
3. Drug/placebo treatment to start

   1. Mild AP Patient is discharged out of the hospital 30 days after diagnosis of mild AP
   2. Moderate Severe or Severe AP Patient is discharged out of hospital Intra-abdominal collections are either resolved on imaging, or are improving and asymptomatic (VAS Pain score ≤3 [with or without pain medication], vomiting ≤once a week, tolerating light diet, and no fever and chills) and do not warrant any intervention (per treating physician)
4. Ability to understand and the willingness to sign a written informed consent document and medical release
5. Willing and able to comply with trial protocol and follow up
6. 2nd AP episode despite correction of the AP etiology (if identified) after the 1st episode as follows i. Patients with biliary pancreatitis who have undergone cholecystectomy, with or without ERCP (if indicated) ii. Patients with hypertriglyceridemia induced pancreatitis who have serum triglyceride levels below 400 while on medication management iii. Patients with medication induced AP developing a 2nd AP episode despite stopping the culprit medication

B- Exclusion Criteria:

1. Age < 18 or > 85 years.
2. Body weight > 200 kg.
3. Ongoing AP (in right clinical situation defined by pain>3, vomiting ≥once a week, fever or chills, not tolerating light diet) or diagnosis of AP in previous 30 days.
4. Diagnosis of chronic pancreatitis, one of the following

   1. Ductal stricture, calcification and/or atrophy, as seen on CT scan/MRI
   2. 5 or more of the 9 EUS criteria used to diagnose CP
5. Known hypersensitivity to Pirfenidone.
6. AST/ALT > 3 times the upper normal limit.
7. Alkaline phosphatase >2.5 times the upper normal limit.
8. Bilirubin higher than upper normal limit.
9. Moderate to severe heart failure and/or coronary heart disease (New York Heart Association (NYHA) Functional Class III/IV).
10. On home oxygen or home mechanical ventilation.
11. Advanced liver disease as defined by Child-Pugh cirrhosis B or C.
12. Paralytic ileus or significant nausea and vomiting preventing administration of light diet.
13. Chronic diarrhea (>6 months, 3 or more stools/day-Clinically not appearing to be steatorrhea [fecal fat if done less than 15 g per day and fecal elastase if done more than 100].Active cancer (on chemotherapy, radiation or treatment of cancer at the time of enrollment) or cancer free <3 years (non-melanoma skin cancer are not a contraindication)
14. Known cancer that is end-stage with ongoing palliative care or for which palliative care is appropriate.
15. Known history of infective hepatitis (Hepatitis B or C)[can enroll if treatment and cure is documented]
16. Ongoing photosensitivity and rash.
17. Known live vaccines or therapeutic infectious agents within one month of admission.
18. Known pregnancy or lactation at the time of admission.
19. Women of childbearing potential who are not on oral or injectable contraceptives or IUDs, and do not consent to adequate contraception while on, and for 90 days after the administration of the drug/placebo.
20. Known to be currently participating in a trial testing any investigational medicinal product or participation in a clinical study involving a medicinal product in the last three months.
21. Problematic pattern of alcohol use or moderate to severe alcohol use disorder (Appendix 2)
22. Substance use disorder (except recreational or medicinal use of marijuana) [if patient underwent and completed a rehab program, has not used substances for at least one year, and has an adequate support system, they may be enrolled]
23. Family or personal history of long QT syndrome (> 500 msec).
24. Strong CYP1A2 inhibitors (e.g., fluvoxamine, enoxacin) or moderate CYP1A2 Inhibitors (e.g., ciprofloxacin).
25. Renal disease with GFR < 30.
26. Any condition other than above that, in the opinion of the investigator, is likely to result in the death of the patient within the next 2 years.
27. Any condition that, in the opinion of the investigator, might be significantly exacerbated by the known side effects associated with the administration of Pirfenidone.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | 6 months
  Development of anticipated or un-anticipated serious adverse events (class 3-4)

SECONDARY OUTCOMES:
Development of Recurrent AP | 2 years
  Cumulative incidence and rate of recurrent attacks of AP over 2 year period following randomization into drug/placebo
Severity of Recurrent Attacks of AP | 2 years
  Classified as mild/moderate/severe
ER Visits | 2 years
  Readmissions and/or ER visits for pain but not AP, over 2 years following randomization into drug/placebo
QOL | 2 years
  SF-12 (0-100, higher score means better physical and mental health functioning)
Patient reported outcomes | 2 years
  Changes in patient reported outcome as measured by PAN-PROMISE score (0-70, with higher score meaning worse symptoms)
Laboratory Marker of Inflammation | 2 years
  Changes in the laboratory markers of inflammation CRP
Laboratory Marker of Inflammation | 2 years
  Changes in the laboratory markers of inflammation IL-10
Laboratory Marker of Inflammation | 2 years
  Changes in the laboratory markers of inflammation TNF-α
Laboratory Marker of Inflammation | 2 years
  Changes in the laboratory markers of inflammation IL-1
Laboratory Marker of Inflammation | 2 years
  Changes in the laboratory markers of inflammation IL-6
Laboratory Marker of Inflammation | 2 years
  Changes in the laboratory markers of inflammation Angiopoietin-2
Development of CP | 2 years
  Fecal Elastase
Development of Chronic Pancreatitis | 2 years
  Development of CP, as evaluated by secretin MRCP at the end of the study
Development of Diabetes | 2 years
  hemoglobin A1C
Development of Diabetes | 2 years
  Fasting blood sugar

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UAB, Birmingham, Alabama
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No